CLINICAL TRIAL: NCT03465254
Title: Effect of Baseline Dengue Serostatus Among Tetravalent Dengue Vaccine CYDTDV (Dengvaxia®) Recipients on Subsequent Virologically Confirmed Dengue in the Philippines
Brief Title: Dengue Serostatus Study in the Philippines
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of the Philippines (Other)
Collaborators: Department of Health, Philippines (Other Government); World Health Organization (Other); Research Institute for Tropical Medicine, Philippines (Other Government); University of North Carolina (Other); La Jolla Institute for Allergy & Immunology (Other); International Vaccine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: UPM REB 2016-435-01
Record Dates: First submitted 2018-03-06; First posted 2018-03-14 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Dengue; Severe Dengue; Dengue Fever; Virologically-confirmed Dengue
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any leftover sera will be used for future studies and stored at UPM-NIH for fifteen (15) years after the end of this study. Future studies using the sera will undergo appropriate ethical reviews as required. After this period, specimens will be destroyed according to local guidelines. Additional consent will be obtained from the parent for storage and future use of these samples. Only the Principal Investigator and designated study personnel will have access to these specimens.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cohort: Recruited members of the cohort are children aged 9-14 years old and eligible to receive the dengue vaccine at the time of the initiation of community-based dengue immunization program of the Department of Health.

SUMMARY:
This is an observational study for 5 years, and aims to determine the risk of developing dengue among Philippine children who are eligible to receive the dengue vaccine during the DOH mass dengue vaccination, by dengue serostatus at baseline.

DETAILED DESCRIPTION:
This is a cohort study that aims to determine the relative risk of developing virologically-confirmed dengue among Philippine children who are eligible to receive dengue vaccine during the DOH Mass Dengue Vaccination. Additionally, it also aims to determine the relative risk of developing severe and/or hospitalized virologically-confirmed dengue among Philippine children who received the Dengue vaccine, describe the epidemiologic trends and characteristics of virologically-confirmed dengue among these children, and assess the performance of simpler tests such as dried blood spots and serum IgG for the assessment of dengue seroprevalence at the population level. We will enroll children who are residents of selected areas in Region 7, Philippines. Children should be eligible to participate in the Department of Health mass dengue vaccination. They will be prospectively venipunctured for baseline dengue serologic status. The blood samples will be stored for serologic testing using neutralization tests and commercial IgG tests. Children in the cohort will be followed up, and those who present with <5 days of fever will be identified and blood drawn for dengue LAMP and RT-PCR.

ELIGIBILITY:
Inclusion criteria:

* Provide signed informed consent and assent (as applicable)
* Be a child belonging to the specified age group and resident of the targeted communities of the DOH dengue mass immunization
* Be eligible to receive dengue vaccine during the DOH dengue mass immunization in 2017

Exclusion criteria:

* Any subject whose parent/guardian refuse to provide informed consent and/or assent
* Children who do not belong to the specified age groups and not residents of the targeted communities
* Children <9 years old
* Children with history of bleeding disorder
* Any subject previously enrolled in a dengue vaccine clinical trial

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children in selected study areas in Region 7, aged 9-14 years old who are considered eligible to be included in the DOH dengue mass vaccination
Sampling Method: Non-Probability Sample
Enrollment: 2996 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
virologically-confirmed dengue (VCD) | 5 years
  The primary outcome measure is virologically confirmed dengue by RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline L. Deen, MD, Principal Investigator — UPM-NIH, Institute of Child Health and Human Development

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lopez AL, Adams C, Ylade M, Jadi R, Daag JV, Molloy CT, Agrupis KA, Kim DR, Silva MW, Yoon IK, White L, Deen J, de Silva AM. Determining dengue virus serostatus by indirect IgG ELISA compared with focus reduction neutralisation test in children in Cebu, Philippines: a prospective population-based study. Lancet Glob Health. 2021 Jan;9(1):e44-e51. doi: 10.1016/S2214-109X(20)30392-2. Epub 2020 Nov 16. PMID 33212030